CLINICAL TRIAL: NCT01867073
Title: A Clinical Pharmacodynamic and Pharmacogenetic Study of OPB-51602 in Patients With Advanced Solid Tumours
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: PG01/04/11
Record Dates: First submitted 2011-05-23; First posted 2013-06-03 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Advanced solid tumours
  Interventions: Other: Biomarker

INTERVENTIONS:
Other: Biomarker

SUMMARY:
OPB-51602 is a novel oral small molecule STAT3 inhibitor developed by Otsuka Pharmaceutical Company, Ltd, and is currently undergoing clinical investigation at the National University Health System (NUHS), Singapore. The proposed correlative pharmacodynamic and pharmacogenetic biomarker study is initiated and funded by the investigators, and will be conducted in conjunction with the extension phase I protocol of OPB-51602 in patients with advanced solid tumours (Study code 266-09-801-01/ DSRB protocol B/09/514). All biomarker and pharmacogenetic samples will be collected, stored and analysed at the local laboratory of the study site (Cancer Science Institute, National University Health System, Singapore, Dr Boon-Cher Goh).

ELIGIBILITY:
Inclusion Criteria:

Advanced Solid Tumor

Exclusion Criteria:

Non advanced solid tumor

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll patients from the extension cohort an ongoing phase I study of OPB51602, to study the tumour response in selected tumour types, as a proof of concept.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-05; Primary Completion 2014-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Inhibition of STAT3 phosphorylation in peripheral mononuclear blood cells (PBMCs)pharmacodynamic effect of OPB-51602 in surrogate tissue. | 1 year
  Analysis

SECONDARY OUTCOMES:
To identify single nucleotide polymorphisms (SNPs) that correlate with OPB-51602 pharmacokinetics and pharmacodynamics | 1 Year
  Analysis

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Yu H, Jove R. The STATs of cancer--new molecular targets come of age. Nat Rev Cancer. 2004 Feb;4(2):97-105. doi: 10.1038/nrc1275. No abstract available. PMID 14964307
- [Background] Buettner R, Mora LB, Jove R. Activated STAT signaling in human tumors provides novel molecular targets for therapeutic intervention. Clin Cancer Res. 2002 Apr;8(4):945-54. PMID 11948098